CLINICAL TRIAL: NCT06120777
Title: Clinical Validation for SpO2 Function of Masimo INVSENSOR00069
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1086
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test Subject (Experimental): All subjects who are enrolled into the test group and participate in data collection have the Masimo INVSENSOR00069.
  Interventions: Device: INVSENSOR00069

INTERVENTIONS:
Device: INVSENSOR00069 — Noninvasive pulse oximeter

SUMMARY:
Assess the accuracy of INVSENSOR00069's peripheral oxygen saturation (SpO2) against contemporaneous measurement from arterial blood gas (ABG) analysis.

ELIGIBILITY:
Inclusion Criteria:

Influenced by study design:

* Subject is 18 to 50 years of age.
* Subject weighs a minimum of 110 lbs.
* Hemoglobin value ≥ 11 g/dL.
* Baseline heart rate ≥ 45 bpm and ≤ 90 bpm.
* Systolic blood pressure ≤ 140 mmHg and ≥ 90 mmHg and diastolic blood pressure ≤ 90 mmHg and ≥ 50 mmHg. If systolic blood pressure is lower than 100 mmHg and/or diastolic blood pressure is lower than 60 mmHg, subject passes an orthostatic blood pressure test.
* CO value ≤ 3.0% FCOHb.
* Subject is comfortable to read and communicate in English*. *This is to ensure the subject can provide informed consent (as study materials are currently available in English only) and can comply with study procedures.

Exclusion Criteria:

Influenced by device warning labels:

* Subjects with a skin condition affecting the digits, where the sensor is applied, which would interfere with the path of light (e.g., psoriasis, vitiligo, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, etc.).
* Subjects with nail polish or acrylic nails on the digits where sensor needs to be applied, who opt not to remove them.
* Subject has hemoglobinopathies or synthesis disorders (e.g., thalassemia, sickle cell disease).
* Subject has a peripheral vascular or vasospastic disease (e.g., Raynaud's disease).

Influenced by study design/environment:

* Subjects who do not pass the health assessment for safe participation in the study procedures.
* Difficulty inserting an intravenous line in the subject's hand or arm and/or an arterial line in the radial artery of the subject's wrist.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Masimo INVSENSOR00069: All subjects who are enrolled into the test group and participate in data collection have the Masimo INVSENSOR00069.
  INVSENSOR00069: Noninvasive pulse oximeter
Period: Overall Study
Arm/Group | Masimo INVSENSOR00069
Started | 89
Completed | 36
Not Completed | 53

BASELINE CHARACTERISTICS:
Arm/Group | Masimo INVSENSOR00069
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 13
  More than one race | 2
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: SpO2 Accuracy of Masimo INVSENSOR00069
Description: The SpO2 accuracy of Masimo INVSENSOR00069 was determined by calculating the accuracy root mean-squared (Arms) difference between the measured values (SpO2) to the reference values (SaO2) in accordance with ISO-80601-2-61.
  Arms= √(∑(i=1 to n) ((SpO2_i-SaO2_i )^2 ))/n.
Time Frame: 1-3 hours
Population: 10 subjects not analyzed due to incorrect sensor 3 subjects not analyzed due to not desaturating to the lowest bin (70-80%)
Measure: Number; unit: % of oxygen saturated hemoglobin
Arm/Group | Masimo INVSENSOR00069
Number analyzed (Participants) | 23
% of oxygen saturated hemoglobin | 1.72

ADVERSE EVENTS:
Time Frame: 1-3 hours
Arm/Group | Masimo INVSENSOR00069
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 9/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Masimo INVSENSOR00069 (N=86)
Dizziness/Lightheadedness (Nervous system disorders) | 5
Nausea (Gastrointestinal disorders) | 1
Hypotension (Cardiac disorders) | 1
Increased heart rate (Cardiac disorders) | 1
Numbness (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT06120777/Prot_SAP_000.pdf